CLINICAL TRIAL: NCT03432013
Title: Targeting Maladaptive Reactivity to Negative Affect in Adolescent Cannabis Users
Brief Title: Affective Management Training for Cannabis Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kate Taylor, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA044350 (NIH)
Record Dates: First submitted 2018-01-30; First posted 2018-02-13 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Cannabis Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUD-CBT (Active Comparator): Standard cognitive behavioral therapy for substance use disorder
  Interventions: Behavioral: SUD-CBT
- CUD-AMT (Experimental): Experimental affective management training for cannabis use disorder specifically
  Interventions: Behavioral: CUD-AMT

INTERVENTIONS:
Behavioral: CUD-AMT — Participants will be trained to manage their negative thoughts and emotions while also receiving treatment for cannabis misuse
  Other Names: Cannabis Use Disorder-Affective Management Treatment
  Arms: CUD-AMT
Behavioral: SUD-CBT — Participants will receive traditional cognitive behavioral therapy for substance use disorder
  Other Names: Substance Use Disorder-Cognitive Behavioral Therapy
  Arms: SUD-CBT

SUMMARY:
Emerging evidence suggests that it is not the negative affect per se but underlying maladaptive cognitive, behavioral, and emotional responses to it that put an individual at risk of pathological substance use. Maladaptive reactivity to negative affect may account for the association between substance-use and emotional disorders and may contribute to poor treatment outcomes for Substance Use Disorder. Thus, teaching adolescents and young adults (herein referred to as "adolescents") skills to manage negative affect may improve therapeutic outcomes of treatment for substance use disorder. Cannabis-use disorder (CUD) among adolescents is a prevalent and growing public health concern. Maladaptive reactivity to negative affect contributes to the maintenance of CUD and accounts for the associations between symptoms of emotional disorders and cannabis use. Still, maladaptive reactivity to negative affect has not yet been targeted in an intervention for CUD. Thus, the overarching aim of this proposal is to develop and pilot test a treatment for CUD that emphasizes the reduction of maladaptive responding to negative affect in adolescents. Participants will be placed in either a standard cognitive behavioral therapy for CUD, or the proposed affective management therapy. The investigators hypothesize that affective management training will yield greater reductions in the participants' use of cannabis, as well as greater improvements to the participants' negative thoughts and emotions, compared to the standard cognitive behavioral therapy.

DETAILED DESCRIPTION:
This project aims to develop and evaluate a behavioral intervention for adolescent cannabis use disorder that emphasizes adaptive responding to negative affective symptoms (e.g., depression, anxiety). Maladaptive cognitive, behavioral, and emotional reactions to negative affect are associated with substance use and substance use problems (including cannabis). Adolescence and young adulthood represents a developmental period in which the regulation of negative emotions is still being developed, as well as a time when cannabis use is prevalent and cannabis use disorders onset. Thus, developing and evaluating cannabis use disorder interventions that emphasize the improvement of responding to negative affect may be particularly important for this developmental period. First, the investigators developed an intervention that weaves skills and strategies for responding adaptively to negative affect, particularly as it relates to high-risk times for cannabis craving and use, into an evidence-based substance use disorder intervention for individuals in late adolescence and early adulthood. After delivering it to a small sample of participants, the investigators will gather feedback to guide refinements to the intervention. After refining the intervention, which will be a 12-session individual treatment, we will conduct the pilot randomized clinical trial. Participants (N = 80) aged 18-25 with cannabis use disorder and elevations in constructs representing maladaptive reactivity to negative affect (i.e., high anxiety sensitivity, low distress tolerance, or facets of emotion dysregulation including high emotional suppression and low cognitive reappraisal ability) will be randomized to receive either: (a) standard cognitive behavioral therapy for adolescent substance use disorders (SUD-CBT) or (b) the novel intervention we develop, affective management training for cannabis use disorders (CUD-AMT). Participants will be assessed at baseline, post-treatment, and a 6-month follow-up assessment on self-report and behavioral indices of the targeted mechanisms, as well as on substance use outcomes (both cannabis-specific and substances more broadly defined). A sub-set of participants (n = 50) will also undergo pre- and post-treatment fMRI assessment to evaluate whether neural indices of emotion regulation are improved to a greater extent in CUD-AMT compared to SUD-CBT. Cannabis use disorder is the most prevalent substance use disorder among adolescents and young adults, and often leads to the use of other substances. Negative affect and disorders associated with high negative affect (i.e., anxiety and unipolar mood disorders) are highly prevalent and associated with significant substance use disorder comorbidity. Targeting a process that is still malleable in late adolescence and young adulthood and that is associated with the maintenance of substance use disorders has the potential to reduce the burden of substance use disorders in this population, thus making a significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

* must be between ages of 18-25; meet diagnostic criteria for cannabis use disorder; score > 1 Standard deviation above the norm on the Positive and Negative Affect Scale-Negative Affect Subscale, and > 1 standard deviation above the norm on either the Anxiety Sensitivity Index, the Distress Tolerance Scale, or the Emotion Regulation Questionnaire; either not on medication or stabilized on medication; fluent in English; and must satisfy usual fMRI criteria.

Exclusion Criteria:

* marked cognitive impairment; moderate to severe suicidality; unstable manic or psychotic symptoms; or primary substance of dependence is not cannabis.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline THC consumption at 3 months and 6 months | baseline, 3 months, and 6 month follow-up
  Urinalysis Toxicology Test primarily assessing levels of THC

SECONDARY OUTCOMES:
Change from baseline in number of cannabis use days at 3 months and 6 months | baseline, 3 months, and 6 month follow-up
  Timeline Followback assesses number of substance use days. At the time of each assessment, the period of time examined is the "past 30 days
Change from baseline additional substance consumption at 3 months and 6 months | baseline, 3 months, and 6 month follow-up
  Urinalysis Toxicology Test used to test for additional substances other than THC
Change in baseline cannabis abuse at 3 months and 6 months | Baseline, 3 months, and 6 month follow-up
  Cannabis Abuse Screening Test assess cannabis-related problems by self-report

CONTACTS AND LOCATIONS:
Overall Officials: Kate Wolitzky-Taylor, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Matrix Institute on Addictions, Los Angeles, California
  - University of California-Los Angeles, Department of Psychiatry and Biobehavioral Sciences, Los Angeles, California